CLINICAL TRIAL: NCT06319300
Title: Efficacy and Safety of the Artificial Intelligence-assisted Insulin Dose Adjustment System for Glycaemic Control in Patients With Type 2 Diabetes Mellitus in General Wards: a Multicentre, Single-blind, Randomised Controlled Study
Brief Title: Artificial Intelligence-assisted Insulin System in Type 2 Diabetes in General Wards
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Shanghai Fifth People's Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20240115023245436
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Type 2
Keywords: diabetes; insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI group (Experimental): AI-assisted insulin dosage adjustment
  Interventions: Device: AI-assisted insulin dose adjustment model
- Doctor group (Active Comparator): doctor adjust insulin
  Interventions: Other: doctor's insulin dose adjustment

INTERVENTIONS:
Device: AI-assisted insulin dose adjustment model — We use an artificial intelligence-assisted insulin dose adjustment system to adjust insulin doses in hospitalised patients
  Other Names: the Artificial Intelligence-assisted Insulin Dose Adjustment System
  Arms: AI group
Other: doctor's insulin dose adjustment — participants' insulin doses are adjusted by doctors
  Arms: Doctor group

SUMMARY:
Our study was a single-blind, randomised, controlled, multicentre study. The study was planned to include 140 patients admitted to the general ward for subcutaneous insulin therapy, who were randomly divided into two groups in the ratio of 1:1, one group with an artificial intelligence assisted insulin dosimetry system to adjust the insulin dose to control their blood glucose, and the other group with a physician instituted insulin dosimetry adjustments to control their blood glucose. The effectiveness and safety of the system was confirmed by comparing the glycaemic control and risk of adverse events between the two groups.

DETAILED DESCRIPTION:
Our study was a single-blind, randomised, controlled, multicentre study. The study was planned to include 140 patients admitted to the general ward for subcutaneous insulin therapy, who were randomly divided into two groups in the ratio of 1:1, one group with an artificial intelligence assisted insulin dosimetry system to adjust the insulin dose to control their blood glucose, and the other group with a physician instituted insulin dosimetry adjustments to control their blood glucose. The effectiveness and safety of the system was confirmed by comparing the glycaemic control and risk of adverse events between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes mellitus > 3 months
* Age≥18 years old
* Receiving glucose-lowering therapy for at least 90 days
* Blood glucose:7.8-22.2 mmol/L
* Length of proposed hospitalisation ≥5 days

Exclusion Criteria:

* Type 1 diabetes mellitus, other special types of diabetes mellitus.
* BG>22.2 mmol/L, or acute complications of diabetes, such as diabetic ketoacidosis, diabetic hyperosmolar state.
* History of severe or repeated hypoglycaemia
* BMI≥45 kg/m2
* Pregnant and lactating women
* Clinically relevant liver disease (established cirrhosis and portal hypertension);
* Presence of severe renal disease (serum creatinine ≥3.0 mg/dL or estimated glomerular filtration rate <30 ml/min/1.73 m2);
* Severe cardiac insufficiency;
* Patients on cortisol-based hormone therapy (equivalent to a prednisone dose >5 mg/day);
* Psychiatric abnormalities or impaired cognitive function;
* Patients with severe oedema, infection, or peripheral blood circulation disorder;
* Patients with severe illness or patients to be transferred to ICU for treatment;
* Surgery of the heart or abdomen that may have a significant impact on the test is planned during hospitalisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-19 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-05-20 (Estimated)

PRIMARY OUTCOMES:
time in target range (3.9-10.0 mmol/L ) | ≥3 days
  Percentage of total time with sensor blood glucose levels in the 3.9-10 mmol/L range

SECONDARY OUTCOMES:
sensor glucose | ≥3 days
  Percentage of total time with sensor blood glucose levels in the range (5.6-10.0mmol/L,10-13.9mmol/L, >13.9mmol/L,<3.0mmol/L, 3.0-3.8mmol/L)
capillary blood sugar | ≥3 days
  pre-breakfast, pre-lunch, pre-dinner, pre-bedtime
hypoglycaemic event | ≥3 days
  capillary blood sugar<3.0 mmol/L
hyperglycaemic event | ≥3 days
  capillary blood sugar>20.0 mmol/L
insulin dosage | ≥3 days
  insulin dosage
satisfaction score of doctors | after intervention
  evaluated by questionnaire.
Length of hospitalisation | ≥3 days
  Length of hospitalisation
Other/Serious Adverse Events | ≥3 days
  Itchy skin, admission to ICU, death, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No